CLINICAL TRIAL: NCT03080415
Title: The Safety and Efficacy of Sofosbuvir & Daclatasvir Combined Therapy for Treatment of Egyptian Children and Adolescents With Chronic Hepatitis C (HCV)-Genotype 4
Brief Title: Treatment of Egyptian Hepatitis C Genotype 4 Infected Children (and Adolescents) With Combined Sofosbuvir & Daclatasvir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yassin Abdelghaffar Charity Center for Liver Disease and Research (Other)
Collaborators: Egyptian Cure Bank (Other); Society of Friends of Liver Patients in the Arab World (SLPAW) (Unknown)
Responsible Party: Principal Investigator, Dr. Tawhida Yassin Abdel Ghaffar, Professor, Yassin Abdelghaffar Charity Center for Liver Disease and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCV SOF T 2017
Record Dates: First submitted 2017-02-22; First posted 2017-03-15 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis C Genotype 4
MeSH Terms: interventions — daclatasvir; Sofosbuvir

STUDY DESIGN:
Intervention Model Description: All of the participants will be receiving combined therapy of sofosbuvir and daclatasvir for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Therapy SOF and DCV (Experimental)
  Interventions: Drug: Combined Therapy SOF and DCV

INTERVENTIONS:
Drug: Combined Therapy SOF and DCV — 1 whole or half tablet sofosbuvir and 1 whole or half tablet daclatasvir per day
  SOF dosage: 400 mg/day for greater than 45 kg weight patients; 200 mg/day for 17 kg to 45 kg patients
  DCV dosage: 60 mg/day for greater than 45 kg weight patients; 30 mg for 17 kg to 45 kg patients
  Other Names: sofosbuvir; daclatasvir

SUMMARY:
This is an open, uncontrolled pilot study of thirty chronic HCV infected patients carried out at Yassin Abdel Ghaffar Charity Center for Liver Disease and Research. The aim of this study is to investigate the safety & efficacy of combined therapy sofosbuvir (SOF) and daclatasvir (DCV) for treating HCV Genotype 4 in children aged 8 to 18. Due to previous positive results in other clinical studies of this drug it is expected that the drug will have high safety and high efficacy. Safety will be measured by checking for adverse effects, while efficacy will be measured by Real-Time Quantitative Polymerase Chain Reaction (qPCR) detecting viral nucleic acids in blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 8-18 years
2. Sex: both sexes
3. Naïve patients, with chronic HCV infection

Exclusion Criteria:

1. Co-infection with Hepatitis B virus (HBV)
2. Other associated chronic liver illness
3. Cirrhotic patients (as indicated by biopsy, fibroscan(F4)
4. Patients with history of hematemesis (non cirrhotic portal hypertension)
5. Patients on drugs known to interact unfavorably with SOF (Amiodarone,..)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | During the 12 weeks of treatment.
  The presence of any adverse effects will be used to characterize this outcome measure.
Sustained Viral Clearance | At Week 12 after end of treatment.
  HCV RNA qPCR will be used to determine if the target of viral clearance has been established. Detection limit of the kit is 12 IU/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Tawhida Y. Abdel Ghaffar, M.D., Principal Investigator — Professor Yassin Abdel Ghaffar Charity Center for Liver Disease and Research
Locations (1):
- Professor Yassin Abdel Ghaffar Charity Center for Liver Disease and Research, Madīnat an Naşr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohd Hanafiah K, Groeger J, Flaxman AD, Wiersma ST. Global epidemiology of hepatitis C virus infection: new estimates of age-specific antibody to HCV seroprevalence. Hepatology. 2013 Apr;57(4):1333-42. doi: 10.1002/hep.26141. Epub 2013 Feb 4. PMID 23172780
- [Background] Wantuck JM, Ahmed A, Nguyen MH. Review article: the epidemiology and therapy of chronic hepatitis C genotypes 4, 5 and 6. Aliment Pharmacol Ther. 2014 Jan;39(2):137-47. doi: 10.1111/apt.12551. Epub 2013 Nov 19. PMID 24251930
- [Background] Messina JP, Humphreys I, Flaxman A, Brown A, Cooke GS, Pybus OG, Barnes E. Global distribution and prevalence of hepatitis C virus genotypes. Hepatology. 2015 Jan;61(1):77-87. doi: 10.1002/hep.27259. Epub 2014 Jul 28. PMID 25069599
- [Background] Gower E, Estes C, Blach S, Razavi-Shearer K, Razavi H. Global epidemiology and genotype distribution of the hepatitis C virus infection. J Hepatol. 2014 Nov;61(1 Suppl):S45-57. doi: 10.1016/j.jhep.2014.07.027. Epub 2014 Jul 30. PMID 25086286
- [Background] Ray SC, Arthur RR, Carella A, Bukh J, Thomas DL. Genetic epidemiology of hepatitis C virus throughout egypt. J Infect Dis. 2000 Sep;182(3):698-707. doi: 10.1086/315786. Epub 2000 Aug 17. PMID 10950762
- [Background] Reker C, Islam KM. Risk factors associated with high prevalence rates of hepatitis C infection in Egypt. Int J Infect Dis. 2014 Aug;25:104-6. doi: 10.1016/j.ijid.2014.02.003. Epub 2014 May 24. PMID 24865321
- [Background] Zahran KM, Badary MS, Agban MN, Abdel Aziz NH. Pattern of hepatitis virus infection among pregnant women and their newborns at the Women's Health Center of Assiut University, Upper Egypt. Int J Gynaecol Obstet. 2010 Nov;111(2):171-4. doi: 10.1016/j.ijgo.2010.06.013. Epub 2010 Aug 12. PMID 20708181
- [Background] El Naghi S, Abdel-Ghaffar TY, El-Karaksy H, Abdel-Aty EF, El-Raziky MS, Allam AA, Helmy H, El-Araby HA, Behairy BE, El-Guindi MA, El-Sebaie H, Abdel-Ghaffar AY, Ehsan NA, El-Hennawy AM, Sira MM. Safety and efficacy of Hansenula-derived PEGylated-interferon alpha-2a and ribavirin combination in chronic hepatitis C Egyptian children. World J Gastroenterol. 2014 Apr 28;20(16):4681-91. doi: 10.3748/wjg.v20.i16.4681. PMID 24782620
- [Background] (CDER) USDoHaHSFaDACfDEaR. Guidance for Industry Chronic Hepatitis C Virus Infection: Developing Direct-Acting Antiviral Drugs for Treatment 2013. Available from: http://www.fda. gov/downloads/drugs/guidancecomplianceregulatoryinformation/ guidances/ucm225333.pdf
- [Background] Peter J, Nelson DR. Optimal interferon-free therapy in treatment-experienced chronic hepatitis C patients. Liver Int. 2015 Jan;35 Suppl 1:65-70. doi: 10.1111/liv.12718. PMID 25529089
- [Background] Papastergiou V, Karatapanis S. Current status and emerging challenges in the treatment of hepatitis C virus genotypes 4 to 6. World J Clin Cases. 2015 Mar 16;3(3):210-20. doi: 10.12998/wjcc.v3.i3.210. PMID 25789294